CLINICAL TRIAL: NCT04106622
Title: Accessory Pathway Antegrade Effective Refractory Period Among Wolff Parkinson White Patients: the Risk in Relation to the Location
Brief Title: Accessory Pathway Antegrade Effective Refractory Period Among WPW Patients: the Risk in Relation to the Location
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Khairy Ibrahim, Principal investigator, Assiut University
Other Study IDs: WPW syndrome
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Wolff-Parkinson-White Syndrome
Keywords: Wolff-Parkinson-White Syndrome
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wolff Parkinson White patients: The investigators will decide the location of the AP by:
  - Invasively: if the patient is subjected to (EPS)
  • There are different locations of AP To assess whether the AP is of high risk or not, for all patients the Antegrade refractory period of the APAERP of the AP will be determined by one of the following ways: ( AERP) is measured during EPS as the shortest cycle length with one-to-one conduction over the AP by incremental atrial stimulation after which the QRS becomes narrow or no conduction occurs due to block of the impulse in the AP. The shortest pre-excited R-R interval (SPERRI) during spontaneous or induced AF.
  The AERP and the risk category of the AP according to its value, will be recorded in relation to the site of the AP determined in every case and compared between different accessory Locations to see whether some of these positions are more liable to be of higher risk or there is no differerence between different positions.
  Interventions: Procedure: electrophysiological study

INTERVENTIONS:
Procedure: electrophysiological study — To assess whether the AP is of high risk or not, for all patients the AERP of the AP will be determined by one of the following ways:
  The cycle length at which abrupt and complete loss of pre-excitation occurs during exercise test. If this didn't happen, the patient will be subjected to invasive electrophysiologic study..
  The Antegrade refractory period of the AP is measured during EPS as the shortest cycle length with one-to-one conduction over the AP by incremental atrial stimulation after which the QRS becomes narrow or no conduction occurs due to block of the impulse in the AP.
  The shortest pre-excited R-R interval during spontaneous or induced AF.

SUMMARY:
To correlate the antegrade effective refractory period of the accessory pathway with its anatomical location in the heart.

To investigate whether the accessory pathway location can predict the high risk nature of the accessory pathway

DETAILED DESCRIPTION:
The Wolf-Parkinson-White (WPW) syndrome is a clinical entity characterized by the presence of ≥1 accessory pathways between the atria and the ventricles pre-disposing patients to arrhythmias. Anterograde conduction through the accessory pathway leads to preexcitation of the ventricles and a delta wave in the ECG. The prevalence of preexcitation in the general population has been estimated to be 1 to 3 in 1000 individuals. Although most asymptomatic patients with pre-excitation have a good prognosis, there is also a lifetime risk of malignant arrhythmias and SCD, estimated to be 0.1 % per patient year.

* More worrisome is the fact that this event can be the first manifestation of the disease in up to 53 % of patients.
* Atrial fibrillation (AF) can be a life-threatening arrhythmia in the WPW syndrome if the AV AP has a short anterograde refractory period (RP), allowing too many atrial impulses to be conducted to the ventricle.
* This will result in very high ventricular rates with possible deterioration into ventricular fibrillation (VF) and sudden death.
* Parameters proved to indicate high risk AP include AP effective refractory period <240 ms, shortest preexcited RR interval <250 ms
* Certain Locations were thought to be associated with higher risk of the accessory pathway like Septal localization which was significantly more frequent in patients with VF when compared with individuals with no VF but the overall number of patients is limited . .

These debatable relations between AP location and its risk stratification was not extensively studied in larger scale studies….

ELIGIBILITY:
1. Inclusion criteria:

   all patients with WPW admitted to Assuit university hospital and subjected to invasive EPS
2. Exclusion criteria:

   1. heart failure
   2. cardiomyopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Wolff Parkinson White patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
the antegrade refractory period during invasive EPS done for the patients | 2 hours
  the values will be correlated to the site of the AP diagnosed be EPS.. according to the previous studies and the current guidelines, if the refractory period is < 250 ms, this is considered a high risk AP

CONTACTS AND LOCATIONS:
Overall Officials: M K Ibrahim, Msc, Principal Investigator — Assiut University; S S Atta, Professor, Study Director — Assiut University; S M Taha, Lecturer, Study Director — Assiut University

REFERENCES:
- Available data/document: Pubmed — https://www.ncbi.nlm.nih.gov/pubmed/